CLINICAL TRIAL: NCT07125638
Title: Long-term Follow-up After OAGB
Status: Completed | Type: Observational
Sponsor: Azienda Sanitaria Locale Napoli 2 Nord (Other)
Responsible Party: Principal Investigator, Francesco Pizza, MD,PhD, Responsible for the Bariatric and Metabolic Surgery unit, Azienda Sanitaria Locale Napoli 2 Nord
Other Study IDs: 0923
Record Dates: First submitted 2025-08-10; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Obesity, Morbid; Obesity, Abdominal; Ona Anastomosis Gastric Bypass; GERD; Bile Reflux Gastritis
MeSH Terms: conditions — Obesity, Morbid; Obesity, Abdominal; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study follows patients who have undergone one-anastomosis gastric bypass (OAGB), a type of weight-loss surgery, to check for changes in the stomach and esophagus over time. All patients have an upper endoscopy before surgery and then again 1, 3, and 5 years later, even if they have no symptoms. The main goal is to see how often problems like bile reflux or ulcers at the surgical join (marginal ulcers) occur. The study also looks at whether patients' symptoms match what is seen during endoscopy.

DETAILED DESCRIPTION:
This study is designed to learn more about changes in the digestive system after one-anastomosis gastric bypass (OAGB), a widely used weight-loss operation. While this surgery is effective for reducing excess weight and improving obesity-related health problems, some people may develop changes in the stomach or esophagus over time, such as bile reflux (backflow of bile into the stomach or esophagus) or marginal ulcers (sores at the site where the stomach is joined to the small intestine).

To better understand how often these problems occur, and whether they cause symptoms, the study follows patients for at least 5 years after surgery. All participants have an upper endoscopy (a camera test that looks at the esophagus, stomach, and the join with the small intestine) before surgery, and then again 1, 3, and 5 years afterwards. These check-ups are done even if the patient feels well, to detect any hidden changes early.

The study also compares what patients report in symptom questionnaires-covering issues like heartburn, regurgitation, or stomach discomfort-with what is actually seen during endoscopy. This will help doctors understand how well symptoms match the real condition of the digestive tract.

By using the same protocol across several specialized bariatric centers, and including all eligible patients, the study aims to provide reliable, long-term data to guide follow-up care after OAGB. The findings could help refine patient monitoring, improve early detection of problems, and identify risk factors that can be addressed to prevent complications.

ELIGIBILITY:
Inclusion Criteria:

* • Age ≥ 18 years.

  * Meets IFSO indications for bariatric surgery (BMI > 40 kg/m², or BMI > 35 kg/m² with obesity-related comorbidities).
  * Candidate for primary one-anastomosis gastric bypass (OAGB).
  * Preoperative upper endoscopy completed as part of standardized work-up.
  * Helicobacter pylori screened preoperatively and (if positive) eradication therapy completed before surgery.
  * Able and willing to attend scheduled postoperative upper endoscopies (at approximately 1, 3, and 5 years) regardless of symptoms.
  * Able to complete patient-reported outcome instruments (GERD-HRQL and abbreviated GSRS).
  * Provided written informed consent.

Ages: 18 Years to 67 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Major postoperative complication within 30 days after OAGB (Clavien-Dindo grade III or IV).
  * Any subsequent abdominal surgery after OAGB (e.g., cholecystectomy, incisional hernia repair) prior to planned endoscopic follow-up.
  * Prior or concomitant revisional bariatric procedure that could impair esophageal motility.
  * Total clinical follow-up shorter than 12 months.
  * Chronic corticosteroid use.
  * Chronic nonsteroidal anti-inflammatory drug (NSAID) use.
  * Preoperative upper endoscopy showing Los Angeles grade ≥ B esophagitis.
  * Preoperative hiatal hernia > 5 cm.
  * Severe, proton-pump-inhibitor-resistant GERD symptoms or advanced lower esophageal sphincter (LES) incompetence preoperatively.
  * Inability or unwillingness to provide informed consent or comply with follow-up.
Sampling Method: Probability Sample
Enrollment: 2368 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Bile Reflux and Marginal Ulcers Assessed by Standardized Endoscopic Follow-up After OAGB | 1 years follow-up
  The primary outcome is the proportion of patients presenting with bile reflux following one-anastomosis gastric bypass (OAGB). Findings are determined through standardized upper gastrointestinal endoscopy performed at 1, 3, and 5 years postoperatively.
  Bile reflux is defined as the presence of visible bile in the gastric pouch or esophagus during endoscopy, with or without associated mucosal changes.
  .
Incidence of Bile Reflux and Marginal Ulcers Assessed by Standardized Endoscopic Follow-up After OAGB | 3 years follow-up
  The primary outcome is the proportion of patients presenting with bile reflux following one-anastomosis gastric bypass (OAGB). Findings are determined through standardized upper gastrointestinal endoscopy performed at 1, 3, and 5 years postoperatively.
  Bile reflux is defined as the presence of visible bile in the gastric pouch or esophagus during endoscopy, with or without associated mucosal changes.
  .
Incidence of Bile Reflux and Marginal Ulcers Assessed by Standardized Endoscopic Follow-up After OAGB | 5 years follow-up
  The primary outcome is the proportion of patients presenting with bile reflux following one-anastomosis gastric bypass (OAGB). Findings are determined through standardized upper gastrointestinal endoscopy performed at 1, 3, and 5 years postoperatively.
  Bile reflux is defined as the presence of visible bile in the gastric pouch or esophagus during endoscopy, with or without associated mucosal changes.
  .
Incidence of Marginal Ulcers After One-Anastomosis Gastric Bypass | 1 years follow-up
  The primary outcome is the proportion of patients developing marginal ulcers following one-anastomosis gastric bypass (OAGB). Marginal ulcers are defined as mucosal ulcerations located at the gastrojejunal anastomosis, confirmed by direct visualization during standardized upper gastrointestinal endoscopy.
  Endoscopy is performed at 1, 3, and 5 years postoperatively, regardless of the presence or absence of symptoms. Lesions are classified according to established endoscopic morphological criteria, and their size, depth, and location are systematically recorded.
Incidence of Marginal Ulcers After One-Anastomosis Gastric Bypass | 3 years follow-up
  The primary outcome is the proportion of patients developing marginal ulcers following one-anastomosis gastric bypass (OAGB). Marginal ulcers are defined as mucosal ulcerations located at the gastrojejunal anastomosis, confirmed by direct visualization during standardized upper gastrointestinal endoscopy.
  Endoscopy is performed at 1, 3, and 5 years postoperatively, regardless of the presence or absence of symptoms. Lesions are classified according to established endoscopic morphological criteria, and their size, depth, and location are systematically recorded.
Incidence of Marginal Ulcers After One-Anastomosis Gastric Bypass | 5 years follow-up
  The primary outcome is the proportion of patients developing marginal ulcers following one-anastomosis gastric bypass (OAGB). Marginal ulcers are defined as mucosal ulcerations located at the gastrojejunal anastomosis, confirmed by direct visualization during standardized upper gastrointestinal endoscopy.
  Endoscopy is performed at 1, 3, and 5 years postoperatively, regardless of the presence or absence of symptoms. Lesions are classified according to established endoscopic morphological criteria, and their size, depth, and location are systematically recorded.

SECONDARY OUTCOMES:
Correlation Between Gastroesophageal Symptoms and Endoscopic Findings After OAGB | 1 year follow-up
  The secondary outcome is the level of agreement between patient-reported gastroesophageal symptoms, assessed using the GERD-Health Related Quality of Life (GERD-HRQL) questionnaire, and objective findings on standardized upper gastrointestinal endoscopy at 1, 3, and 5 years after one-anastomosis gastric bypass (OAGB). Concordance is measured using the Cohen's kappa statistic, with symptoms recorded as present/absent and endoscopic lesions classified according to the Los Angeles grading system for esophagitis and established criteria for gastritis and ulcer disease.
Correlation Between Gastroesophageal Symptoms and Endoscopic Findings After OAGB | 3 year follow-up
  The secondary outcome is the level of agreement between patient-reported gastroesophageal symptoms, assessed using the GERD-Health Related Quality of Life (GERD-HRQL) questionnaire, and objective findings on standardized upper gastrointestinal endoscopy at 1, 3, and 5 years after one-anastomosis gastric bypass (OAGB). Concordance is measured using the Cohen's kappa statistic, with symptoms recorded as present/absent and endoscopic lesions classified according to the Los Angeles grading system for esophagitis and established criteria for gastritis and ulcer disease.
Correlation Between Gastroesophageal Symptoms and Endoscopic Findings After OAGB | 5 year follow-up
  The secondary outcome is the level of agreement between patient-reported gastroesophageal symptoms, assessed using the GERD-Health Related Quality of Life (GERD-HRQL) questionnaire, and objective findings on standardized upper gastrointestinal endoscopy at 1, 3, and 5 years after one-anastomosis gastric bypass (OAGB). Concordance is measured using the Cohen's kappa statistic, with symptoms recorded as present/absent and endoscopic lesions classified according to the Los Angeles grading system for esophagitis and established criteria for gastritis and ulcer disease.

CONTACTS AND LOCATIONS:
Overall Officials: francesco pizza, PhD, Principal Investigator — Azienda Sanitaria Locale Napoli 2 Nord
Locations (1):
- Azienda Sanitaria Locale Napoli 2 Nord - U.O.C. Chirurgia Generale, P.O. "Anna Rizzoli", Lacco Ameno, Naples, Italy, Naples, naples, Italy